CLINICAL TRIAL: NCT00217620
Title: Phase II Trial of BAY-9006 (NSC #724772) in Advanced Soft Tissue Sarcomas
Brief Title: S0505 Sorafenib in Treating Patients With Advanced Soft Tissue Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03063; S0505 (Other: SWOG); U10CA032102 (NIH); CDR0000442404 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2013-01

CONDITIONS: Sarcoma
Keywords: adult angiosarcoma; adult leiomyosarcoma; adult liposarcoma; adult malignant hemangiopericytoma; recurrent adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma; Leiomyosarcoma; Liposarcoma; Hemangiopericytoma, Malignant | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sorafenib (Experimental): sorafenib
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — 800 mg per day, daily until progression
  Other Names: BAY 43-9006

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sorafenib works in treating patients with advanced soft tissue sarcomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate (confirmed, complete, and partial) in patients with advanced soft tissue sarcomas treated with sorafenib.
* Determine the 4-month progression-free survival rate in patients treated with this drug.
* Determine the frequency and severity of adverse events in patients treated with this drug.

OTHER OBJECTIVES (if funding permits):

* Correlate, preliminarily, a decrease in standard uptake variable (SUV) of target lesions by positron-emission tomography scan at 4 weeks with response in patients treated with this drug.
* Correlate, preliminarily, the phosphorylation status of KIT, PDGFR, VEGFR, and the raf/mek/erk pathway with response in patients treated with this drug.
* Correlate, preliminarily, the most common B-raf kinase mutation with response in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to histology (leiomyosarcoma vs liposarcoma vs angiosarcoma, hemangiosarcoma, or hemangiopericytoma).

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 8 weeks until disease progression and then every 6 months for 2 years and annually for up to 3 years.

PROJECTED ACCRUAL: A total of 45-75 patients (15-25 per stratum) will be accrued for this study within 15-38 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma of 1 of the following histologies:

  * Angiosarcoma, cutaneous or visceral
  * Malignant hemangiosarcoma
  * Malignant hemangiopericytoma
  * Grade 3-4 leiomyosarcoma
  * Grade 3-4 liposarcoma
* Must have evidence of unresectable residual disease, metastatic disease, or recurrent disease by radiography
* Measurable disease by x-ray, scans, or physical examination
* Archived paraffin-embedded tumor sections available
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if due to liver metastases)
* Bilirubin normal (≤ 2.5 times ULN if due to liver metastases)
* PT, PTT, and INR normal

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No history of thromboembolic disease
* No uncontrolled hypertension

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to swallow oral medication
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 28 days since prior chemotherapy (42 days for carmustine or mitomycin) and recovered
* Prior adjuvant chemotherapy allowed
* No more than 1 prior chemotherapy regimen for metastatic disease

Endocrine therapy

* Not specified

Radiotherapy

* At least 28 days since prior radiotherapy and recovered

  * Must have evidence of disease progression within, or measurable disease outside of, the radiation field after completion of radiotherapy

Surgery

* At least 28 days since prior major surgery and recovered

Other

* No prior sorafenib
* No prior inhibitor of VEGFR or MAPK pathway
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent therapeutic anticoagulation
* No concurrent administration of any of the following medications:

  * Rifampin
  * Hypericum perforatum (St. John's wort)
  * Cytochrome P450 enzyme-inducing antiepileptic drugs, including any of the following:

    * Phenytoin
    * Carbamazepine
    * Phenobarbital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, MD, Study Chair — Fox Chase Cancer Center; George D. Demetri, MD, Study Chair — Dana-Farber Cancer Institute
Locations (184):
- United States (184):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Sutter Solano Medical Center, Vallejo, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - Bettendorf, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA at Maplewood Cancer Center, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest Virginia Regional Cancer Center, Norton, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Ryan CW, von Mehren M, Rankin CJ, et al.: Phase II intergroup study of sorafenib (S) in advanced soft tissue arcomas (STS): SWOG 0505. [Abstract] J Clin Oncol 26 (Suppl 15): A-10532, 2008.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib (BAY 43-9006): Sorafenib (BAY 43-9006) 800 mg per day divided into two equal doses of 400 mg by mouth (PO). Patients received the drug continuously on a daily basis until progression; each cycle is 28 days. All eligible patients who received treatment were included in baseline measures.
Period: Overall Study
Arm/Group | Sorafenib (BAY 43-9006)
Started | 51
Eligible | 38
Eligible and Began Protocol Therapy | 37
Completed | 0
Not Completed | 51
Not completed — Adverse Event | 2
Not completed — Progression | 31
Not completed — Not Protocol Specified | 4
Not completed — Ineligible | 13
Not completed — Never received treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib (BAY 43-9006)
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 62.7 [24.0 to 88.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 15
Race/Ethnicity, Customized [Number; unit: participants]
  White | 33
  Black | 3
  Pacific Islander | 1
Histology [Number; unit: participants]
  Leiomyosarcoma | 19
  Liposarcoma | 10
  Soft Tissue Sarcoma of Vascular Derivation | 8
Performance Status [Number; unit: participants] — Performance status is graded according to the Zubrod Performance Status Scale. Patients with a performance status of 0 are fully active, able to carry on all pre-disease performance without restriction. Patients with a performance status of 1 are restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  participants
    0 | 15
    1 | 22

OUTCOME MEASURES:

1. Secondary Outcome: Four-month Progression-free Survival Rate
Time Frame: 0 - 4 months
Population: Eligible patients who had received any treatment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Leiomyosarcoma; Liposarcoma; Vascular Sarcomas; Total: Sorafenib (BAY 43-9006) 800 mg per day divided into two equal doses of 400 mg by mouth (PO). Patients received the drug continuously on a daily basis until progression; each cycle is 28 days. All eligible patients who received treatment were included in baseline measures.
Arm/Group | Leiomyosarcoma | Liposarcoma | Vascular Sarcomas | Total
Number analyzed (Participants) | 19 | 10 | 8 | 37
percentage of participants | 42 [20 to 64] | 30 [2 to 58] | 63 [29 to 96] | 43 [27 to 59]

2. Primary Outcome: Objective Response (Confirmed, Complete and Partial)
Description: Partial response (PR) is greater than or equal to 30% decrease under baseline of sum of longest diameters of all target measurable lesions; No unequivocal progression of non-measurable disease; No new lesions. Unconfirmed PR is one objective status of PR documented before progression or symptomatic deterioration. Stable disease does not qualify for CR, PR, Progression or Symptomatic Deterioration. Progressive disease is any one or more of the following: 20% increase in sum of longest diameters of target measurable lesions over smallest sum observed; unequivocal progression of non-measurable disease; appearance of any new lesion/site; death due to disease without prior documentation of progression and without symptomatic deterioration. Assessment inadequate is progression or symptomatic deterioration has not been documented, and one or more target measurable lesions have not been assessed or inconsistent assessment methods were used.
Time Frame: Assessment performed every eight weeks until progression.
Population: Eligible patients who had received any treatment were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Leiomyosarcoma | Liposarcoma | Vascular Sarcomas
Number analyzed (Participants) | 19 | 10 | 8
participants
  Unconfirmed PR | 1 | 0 | 1
  Stable disease/no response | 8 | 2 | 5
  Progressive disease | 9 | 6 | 1
  Assessment inadequate | 1 | 2 | 1

3. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 3.0. For each patient, worst grade of each event type is reported. Grade 3 - Severe, Grade 4 - Life-threatening, Grade 5 - Fatal. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Patients were assessed for adverse events two weeks after starting protocol treatment and then after every cycle of treatment (1 cycle = 28 days) for the duration of protocol treatment.
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Sorafenib (BAY 43-9006)
Number analyzed (Participants) | 37
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1
  AST, SGOT | 1
  Alkaline phosphatase | 1
  Amylase | 1
  Bilirubin (hyperbilirubinemia) | 1
  Constipation | 1
  Diarrhea | 4
  Fatigue (asthenia, lethargy, malaise) | 2
  Hemoglobin | 1
  Hypertension | 2
  Lipase | 6
  Nausea | 1
  Pain - Abdomen NOS | 1
  Pancreatitis | 1
  Platelets | 1
  Potassium, serum-low (hypokalemia) | 2
  Rash/desquamation | 2
  Rash: hand-foot skin reaction | 4
  Sodium, serum-low (hyponatremia) | 2
  Vomiting | 1

ADVERSE EVENTS:
Time Frame: Patients assessed for adverse events 2 weeks after starting treatment and then after every cycle (28 days) for the duration of protocol treatment. Assessments continued until resolution of any adverse events up to 5 years after registration.
Arm/Group | Sorafenib (BAY 43-9006)
Serious Adverse Events (participants affected / at risk) | 10/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (BAY 43-9006) (N=37)
Hemoglobin (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Hemorrhage, GI - Colon (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 3
Pancreatitis (Gastrointestinal disorders) | 1
Pain - Chest/thorax NOS (General disorders) | 1
AST, SGOT (Investigations) | 1
Amylase (Investigations) | 1
Lipase (Investigations) | 2
Platelets (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Mental status (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Obstruction, GU - Ureter (Renal and urinary disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (BAY 43-9006) (N=37)
Blood/Bone Marrow-Other (Specify) (Blood and lymphatic system disorders) | 6
Hemoglobin (Blood and lymphatic system disorders) | 8
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 19
Flatulence (Gastrointestinal disorders) | 4
Heartburn/dyspepsia (Gastrointestinal disorders) | 4
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 14
Pain - Abdomen NOS (Gastrointestinal disorders) | 8
Pain - Oral cavity (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 8
Edema: limb (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 23
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 4
Allergic reaction/hypersensitivity (Immune system disorders) | 2
Infection-Other (Specify) (Infections and infestations) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 8
AST, SGOT (Investigations) | 13
Alkaline phosphatase (Investigations) | 11
Amylase (Investigations) | 7
Bilirubin (hyperbilirubinemia) (Investigations) | 3
Creatinine (Investigations) | 7
Leukocytes (total WBC) (Investigations) | 3
Lipase (Investigations) | 9
Lymphopenia (Investigations) | 6
Metabolic/Laboratory-Other (Specify) (Investigations) | 4
PTT (Partial thromboplastin time) (Investigations) | 3
Platelets (Investigations) | 2
Weight loss (Investigations) | 10
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 15
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 10
Pain - Back (Musculoskeletal and connective tissue disorders) | 4
Pain - Bone (Musculoskeletal and connective tissue disorders) | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 5
Pain - Joint (Musculoskeletal and connective tissue disorders) | 7
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 5
Pain - Head/headache (Nervous system disorders) | 5
Taste alteration (dysgeusia) (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 4
Mood alteration - anxiety (Psychiatric disorders) | 2
Renal/Genitourinary-Other (Specify) (Renal and urinary disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 3
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 2
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 7
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 14
Pain - Scalp (Skin and subcutaneous tissue disorders) | 5
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 14
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 21
Flushing (Vascular disorders) | 4
Hypertension (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less